CLINICAL TRIAL: NCT03718403
Title: Effect of Theophylline in Pseudohypoparathyroidism
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Amita Sharma, Medical Director, Division of Pediatric Nephrology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Theophylline in PHP
Record Dates: First submitted 2017-09-08; First posted 2018-10-24 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: PHP Ia; PHP IB; Php1C
Keywords: PHP
MeSH Terms: conditions — Pseudohypoparathyroidism; Pseudohypoparathyroidism Type 1C | interventions — Theophylline

STUDY DESIGN:
Intervention Model Description: Open label intervention study, off label use of theophylline
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Single arm open labeled intervention study (Experimental): Subjects with PHP will be given theophylline to decrease the end organ resistance by increasing levels of cAMP, a second messenger. Theophylline will be dosed twice a day for a period of 52 weeks.
  Interventions: Drug: Theophylline

INTERVENTIONS:
Drug: Theophylline — Theophylline will be given to maintain a peak level between 10-15 mcg/mL

SUMMARY:
The study evaluates the effect of theophylline in 100 subjects with Pseudohypoparathyroidism.

DETAILED DESCRIPTION:
It is an open label intervention study for the off-label use of theophylline in psuedohypoparathyroidism (PHP).Theophylline is a is non-specific phosphodiesterase inhibitor which increases the levels of secondary messenger,cAMP. PHP patients have end organ resistance to hormones involving cAMP signaling. Thus, theophylline has a potential to abrogate hormone resistance. Also, it may have a role in bone maturation, neurocognition and metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with known diagnosis of PHP1A and PHP1B
* Age >5 years

Exclusion Criteria:

* • Significant kidney disease, i.e. any CKD stage

  * Hypercalciuria
  * Kidney stones
  * Severe Heart disease
  * Uncontrolled seizure disorder
  * Peptic ulcer
  * Liver dysfunction
  * Bleeding disorder
  * Allergy to theophylline preparation
  * Muscle disorder
  * Infection
  * Any neurologic disease
  * Chronic drugs interacting with theophylline

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-11-11 (Actual); Primary Completion 2030-04-10 (Estimated); Study Completion 2032-04-10 (Estimated)

PRIMARY OUTCOMES:
Effect of Theophylline on Bone Age in PHP | 52 weeks
  Change in Bone age ( in years and months) before and after theophylline administration for 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: AMITA SHARMA, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States